CLINICAL TRIAL: NCT01885871
Title: Safety and Efficacy of Cutera Picosecond Q-Switched Nd:YAG Laser in the Treatment of Solar Lentigines
Brief Title: Laser Removal of Age (Sun) Spots on Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-13-LPS03; C-13-LPS03 (Other: Cutera)
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2015-10

CONDITIONS: Solar Lentigines
Keywords: Sun; Age; Spot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Picosecond QS Nd:YAG Laser (Experimental): Laser Treatment with Investigational Device
  Interventions: Device: Picosecond QS Nd:YAG Laser

INTERVENTIONS:
Device: Picosecond QS Nd:YAG Laser — Up to 2 laser treatments delivered 6 weeks apart
  Other Names: Cutera

SUMMARY:
The purpose of this study is to determine whether picosecond laser is effective in the treatment of age (sun) spots.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of Cutera Picosecond Q-Switched Nd:YAG 1064 and/or 532 nm laser in the treatment of benign pigmented lesions on the hands.

ELIGIBILITY:
Inclusion Criteria:

* Females or Males, 18 to 60 years of age (inclusive).
* Fitzpatrick Skin Type I - III (Appendix 2).
* Clinical diagnosis of benign solar lentigines of the hands.
* Presence of at least 5 lesions in the treatment area in diameters ranging from 1 to 8 mm.
* Has not used any prescription or over the counter topical creams (e.g., hydroquinone, and/or retinoids and/or corticosteroids) used in the treatment of pigmentation in the treatment area within the last 4 weeks.
* Willing to refrain from using any prescription or over the counter topical creams used for the treatment of pigmentation (e.g., hydroquinone, and/or retinoids and/or corticosteroids) in the treatment area during the study period.
* Must be able to read, understand and sign the Informed Consent Form.
* Willing and able to adhere to the treatment and follow-up schedule and before and after treatment care instructions.
* Willing to protect and/or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher in the treatment area starting up to 4 weeks before the treatment, every day for the duration of the study, including the follow-up period
* Willing to have digital photographs taken of the treatment area
* Agree not to undergo any other procedure(s) for the treatment of solar lentigines during the study.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at last 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

* Participation in a study of another device of drug within 6 months prior to enrollment or during the study.
* Prior treatment of solar lentigines of the hands, e.g., with Q-Switched laser, IPL, Chemical peel, cryotherapy within 6 months of study participation.
* Having pre-malignant or malignant lesions (e.g., pigmented actinic keratosis, lentigo maligna [12], lentigo maligna melanoma), or history of a pre-malignant or malignant lesion in the treatment area.
* Subject shows signs of actinic bronzing or recent tanning in the treatment area, and unable/unlikely to refrain from tanning during the study.
* Skin abnormalities in the treatment area, e.g., cuts, scrapes, wounds, scars, large moles.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* History of immunosuppression/immune deficiency disorders or currently using immunosuppression medications.
* History of vitiligo or psoriasis.
* History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light, such as tetracycline.
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Current smoker or history of smoking within 2 years of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.
* History of allergy to topical antibiotics.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Moldre, NP, Principal Investigator — Cutera Inc.
Locations (1):
- Cutera Research Center, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Picosecond Q-Switched Nd:YAG 1064/532 nm Laser: Picosecond Q-Switched Nd:YAG 1064/532 nm Laser: Up to 2 laser treatments delivered 6 weeks apart
Period: Overall Study
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 52 [41 to 67]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Median VAS Improvement Score as Assessed by Blinded Physician Reviewers
Description: Improvement (clearing) in solar lentigines as assessed by blinded physician reviewers using a VAS 4 point scale 0-3 where 0=no change and 3=Very much improved.
Time Frame: 12 weeks post- final treatment
Population: Based on blinded photographic assessments of 20 subjects. Scores >/=1 indicate clearing.
Measure: Median (95% Confidence Interval); unit: units on a scale
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Number analyzed (Participants) | 20
units on a scale | 1.5 [1.25 to 2]
Statistical Analysis 1: Comparison: Picosecond Q-Switched Nd:YAG 1064/532 nm Laser; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percent of Participants With Improvement Score >/=1
Description: Improvement (clearing) in solar lentigines as assessed by participant using a 4-point VAS 0-3 scale where 0=no change and 3=very much improved. Scores >/=1 indicate improvement.
Time Frame: 12 weeks post- final treatment
Measure: Number; unit: percent of participants
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Number analyzed (Participants) | 20
percent of participants | 90

3. Secondary Outcome: Percent of Participants Satisfied With Improvement (Clearing) in Solar Lentigines
Description: Level of Satisfaction with Improvement (clearing) in solar lentigines as assessed by participants, as measured by spot Improvement: 3=Very Much Improved, 2=Much Improved, 1=Improved, and 0=No Change.
Time Frame: 12 weeks post- final treatment
Population: Based on subject questionnaires, 90% of subjects reported improvement (clearing) in benign pigmented lesions at 12 weeks post- final treatment. Scores > or =1 indicate improvement.
Measure: Number; unit: percent of participants
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Number analyzed (Participants) | 20
percent of participants | 95

4. Secondary Outcome: Mean Pain Score Associated With Laser Treatments
Description: Subjects graded the level of pain associated with each laser treatment, using a 0-10 scale where 0=no pain and 10=worse possible pain, then averaged to get the mean across the treatments.
Time Frame: During treatments
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Number analyzed (Participants) | 20
units on a scale | 2.0 [1.0 to 5.0]

5. Secondary Outcome: Percent of Subjects With Post-treatment Adverse Event
Time Frame: During study duration 0-6 months.
Measure: Number; unit: percent of participants
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Number analyzed (Participants) | 20
percent of participants
  Erythema (redness) | 100
  Edema (swelling) | 100
  Crusting (scabbing) | 100
  Purpura (bruising) | 65
  Blisters | 15
  Eczema | 5

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected immediately post treatment, 3 days and 14 days after treatment as well as 6, 12, and 24 weeks.
Arm/Group | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Picosecond Q-Switched Nd:YAG 1064/532 nm Laser (N=20)
Edema (swelling) (Skin and subcutaneous tissue disorders) | 20 (20)
Erythema (Redness) (Skin and subcutaneous tissue disorders) | 20 (20)
Purpura (Bruising) (Skin and subcutaneous tissue disorders) | 13 (13)
Blisters (Skin and subcutaneous tissue disorders) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes